CLINICAL TRIAL: NCT00767637
Title: Open Label, Non-controlled Long-term Treatment on BAY77-1931 (Lanthanum Carbonate) to Measure Lanthanum Concentrations in Bone in Patients With Hyperphosphatemia Receiving Dialysis
Brief Title: Long-term Treatment on BAY77-1931 (Lanthanum Carbonate) to Measure Lanthanum Concentrations in Bone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11810; Fosrenol (Other: Company Internal)
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Hyperphosphatemia; Dialysis
MeSH Terms: conditions — Hyperphosphatemia | interventions — lanthanum carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Lanthanum Carbonate (BAY77-1931)

INTERVENTIONS:
Drug: Lanthanum Carbonate (BAY77-1931) — BAY77-1931 750mg, in the morning, day and evening

SUMMARY:
To measure lanthanum concentrations in bone in patients with hyperphosphatemia receiving dialysis

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing dialysis or plan to start dialysis before the initial administration of the study medication

Exclusion Criteria:

* Patients with severe hypocalcemia (adjusted serum calcium level of <7.5 mg/dL)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2005-06; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Changes in pre-dialysis serum phosphate levels | Every 2 weeks

SECONDARY OUTCOMES:
Achievement rate of the target predialysis serum phosphate levels (3.5 mg/dL and 5.5 mg/dL) | Every 2 weeks
Changes in corrected serum calcium level | Every 2 weeks
Changes in the product of serum calcium and phosphate | Every 2 weeks
Changes in serum intact-PHT levels | Every 2 weeks
Changes in bone metabolism markers | Every 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Japan (2):
  - Isesaki, Gunma
  - Yonago, Tottori

REFERENCES:
- [Derived] Shigematsu T, Tokumoto A, Nakaoka A, Arisaka H. Effect of lanthanum carbonate treatment on bone in Japanese dialysis patients with hyperphosphatemia. Ther Apher Dial. 2011 Apr;15(2):176-84. doi: 10.1111/j.1744-9987.2010.00898.x. PMID 21426511